CLINICAL TRIAL: NCT05196061
Title: Human Skin and Gut Mycobiome and Bacteriome Comprehensive Registry
Status: Recruiting | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Mahmoiud A. Ghannoum, Principal Investigator, University Hospitals Cleveland Medical Center
Other Study IDs: STUDY20191290
Record Dates: First submitted 2021-12-15; First posted 2022-01-19 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Surveys and Questionnaires; Mouthwashes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Questionnaire — Subjects will be asked to complete a questionnaire. The questionnaire will garner demographic data, medical history, medication and supplement history, gut-specific, skin-specific questions; etc. The complete questionnaire is provided with this submission for review. Demographic data includes:
  1. Age
  2. Sex
  3. Race
  4. Ethnicity
Other: Stool sample — Stool samples will be collected using a specific kit consisting of a ready-to-use package, including a user guide. When stool samples are collected, they will be immediately placed in previously prepared Fast prep tubes (MP, Cat# 5076-200-34340) containing 500 μL glass beads (Sigma-Aldrich G8772-100g) and 1 mL ASL™ lysis buffer (Qiagen DNA Extraction Kit) and transported to the laboratory where assays will be conducted. Samples will be kept in a - 20 degree Celsius freezer until they are analyzed.
Other: Skin swab — Skin swabbing is a safe, non-invasive method to sample microbiota on human skin. Areas to be swabbed: Right upper back, Non-dominant ventral forearm or Most representative lesion
Other: Oral rinse — Briefly, 20-25 ml saline will be provided in separately labelled blue capped 50-mL Falcon™ centrifuge tubes (Fisher Scientifics Co.). Each subject will be asked to swish and gargled the saline from the tube into their mouth for 2 minutes and expectorate the rinse into the tube. The tubes will be closed tightly and stored in -80 C until sequencing can be completed. Prior to use, all the tubes with oral wash samples will be completely thawed on ice, then centrifuged at 4000 rpm for 15 minutes and 20-25 ml supernatant transferred into fresh 50-mL centrifuge tubes. The pellet left in each tube will be used to extract DNA for microbiome studies

SUMMARY:
Bacterial and fungal microbiota will be different between individual body sites; however, particular microbiome profiles both whole-body and site-specific will be unique to volunteers with a given parameter such as medical diagnosis, diet, medications taken, geographical area; etc.

DETAILED DESCRIPTION:
Specific aims:

1. Identify and characterize whole-body and site-specific microbiome profiles.
2. Identify phenotypic microbiome profiles unique to individual parameters such as demographics, medical diagnoses, diet; etc.
3. Perform bacterial-bacterial, fungal-fungal and bacterial-fungal correlation analysis to identify potential synergistic and antagonistic species within these unique profiles.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving informed consent.
* Able and willing to complete all required specified study procedures

Exclusion Criteria:

* Antibiotic or antifungal use whether topical or systemic in the past 2 or 4 weeks, respectively.
* Unable and/or unwilling to complete all required study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers will be age 18 years or older and capable of giving informed consent and able and willing to complete all required study specified procedures
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
whole-body and site-specific microbiome profiles | through study completion, an average of 10 year
  Identify and characterize whole-body and site-specific microbiome profiles.
Phenotypic microbiome profiles unique to individual parameters | through study completion, an average of 10 year
  Identify phenotypic microbiome profiles unique to individual parameters such as demographics, medical diagnoses, diet; etc.
bacterial-bacterial, fungal-fungal and bacterial-fungal correlation analysis | through study completion, an average of 10 year
  Perform bacterial-bacterial, fungal-fungal and bacterial-fungal correlation analysis to identify potential synergistic and antagonistic species within these unique profiles.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
results will not be shared with other researchers

REFERENCES:
- [Background] Muszer M, Noszczynska M, Kasperkiewicz K, Skurnik M. Human Microbiome: When a Friend Becomes an Enemy. Arch Immunol Ther Exp (Warsz). 2015 Aug;63(4):287-98. doi: 10.1007/s00005-015-0332-3. Epub 2015 Feb 15. PMID 25682593
- [Background] Ackerman J. The ultimate social network. Sci Am. 2012 Jun;306(6):36-43. doi: 10.1038/scientificamerican0612-36. No abstract available. PMID 22649992
- [Background] Proctor LM. The Human Microbiome Project in 2011 and beyond. Cell Host Microbe. 2011 Oct 20;10(4):287-91. doi: 10.1016/j.chom.2011.10.001. PMID 22018227
- [Background] Ursell LK, Metcalf JL, Parfrey LW, Knight R. Defining the human microbiome. Nutr Rev. 2012 Aug;70 Suppl 1(Suppl 1):S38-44. doi: 10.1111/j.1753-4887.2012.00493.x. PMID 22861806
- [Background] Dave M, Higgins PD, Middha S, Rioux KP. The human gut microbiome: current knowledge, challenges, and future directions. Transl Res. 2012 Oct;160(4):246-57. doi: 10.1016/j.trsl.2012.05.003. Epub 2012 Jun 7. PMID 22683238
- [Background] Grice EA, Kong HH, Conlan S, Deming CB, Davis J, Young AC; NISC Comparative Sequencing Program; Bouffard GG, Blakesley RW, Murray PR, Green ED, Turner ML, Segre JA. Topographical and temporal diversity of the human skin microbiome. Science. 2009 May 29;324(5931):1190-2. doi: 10.1126/science.1171700. PMID 19478181
- [Background] Grice EA, Segre JA. The skin microbiome. Nat Rev Microbiol. 2011 Apr;9(4):244-53. doi: 10.1038/nrmicro2537. PMID 21407241
- [Background] Mukherjee PK, Chandra J, Retuerto M, Tatsuoka C, Ghannoum MA, McComsey GA. Dysbiosis in the oral bacterial and fungal microbiome of HIV-infected subjects is associated with clinical and immunologic variables of HIV infection. PLoS One. 2018 Jul 11;13(7):e0200285. doi: 10.1371/journal.pone.0200285. eCollection 2018. PMID 29995962